CLINICAL TRIAL: NCT01136733
Title: An Open-Label, Multicenter, Phase 1b/2 Study of E7080 Alone, and in Combination With Everolimus in Subjects With Unresectable Advanced or Metastatic Renal Cell Carcinoma Following One Prior VEGF-Targeted Treatment
Brief Title: A Study of E7080 Alone, and in Combination With Everolimus in Subjects With Unresectable Advanced or Metastatic Renal Cell Carcinoma Following One Prior Vascular Endothelial Growth Factor (VEGF)-Targeted Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-205
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Unresectable advanced or metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib; Everolimus

ARMS (3):
- Lenvatinib (Experimental)
  Interventions: Drug: Lenvatinib
- Lenvatinib plus Everolimus (Experimental)
  Interventions: Drug: Lenvatinib; Drug: Everolimus
- Everolimus (Active Comparator)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Lenvatinib — taken orally, once a day
  Other Names: E7080, Lenvima, Kisplyx
  Arms: Lenvatinib; Lenvatinib plus Everolimus
Drug: Everolimus — taken orally, once a day
  Other Names: Afinitor
  Arms: Everolimus; Lenvatinib plus Everolimus

SUMMARY:
This is an open-label, multicenter, Phase 1b/2 study of lenvatinib alone and in combination with everolimus in subjects with unresectable advanced or metastatic renal cell carcinoma following one prior VEGF-targeted treatment.

ELIGIBILITY:
Select Inclusion Criteria:

* Histologically confirmed diagnosis of renal cell carcinoma.
* Phase 2: Histological or cytological confirmation of predominant clear cell renal cell carcinoma (RCC) (original tissue diagnosis of RCC is acceptable).
* Documented evidence of unresectable advanced or metastatic RCC. Phase 2: Radiographic evidence of disease progression according to modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Phase 2: One prior vascular endothelial growth factor (VEGF)-targeted treatment (for example, but not limited to, sunitinib, sorafenib, pazopanib, bevacizumab, axitinib, vatalanib, AV951/tivozanib) for unresectable advanced or metastatic RCC.
* Phase 2: Measurable disease meeting the following criteria: a.) at least 1 lesion of greater than or equal to 1.5 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short axis diameter for a lymph node which is serially measurable according to Modified RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI) or photography. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Screening Visit.

Select Exclusion Criteria:

Phase 1b or Phase 2 specific per below:

* Phase 1b only: Subjects with untreated or unstable metastasis to the central nervous system (CNS) are excluded. Subjects who have completed local therapy and have discontinued the use of steroids for this indication at least 4 weeks prior to commencing treatment and in whom stability has been proven by at least 2 CT or MRI scans obtained at least 4 weeks apart are eligible for Phase 1b only. Phase 2 only: Subjects with CNS (e.g., brain or leptomeningeal) metastasis are excluded.
* Phase 2 only: More than one prior VEGF-targeted treatment for unresectable advanced or metastatic RCC.

Phase 1b or Phase 2 specific per below:

* Phase 1b only: Prior exposure to lenvatinib. Phase 2 only: Prior exposure to lenvatinib or mammalian target of rapamycin (mTOR) inhibitor.
* Subjects should not have received any anticancer treatment within 21 days or any investigational agent within 30 days prior to the first dose of study drug and should have recovered from any toxicity related to previous anticancer treatment. Major surgery within 3 weeks prior to the first dose of study drug.
* Subjects having greater than 1+ proteinuria on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria.
* Subjects with urine protein greater than or equal to 1 g/24 hours will be ineligible. Uncontrolled diabetes as defined by fasting serum glucose at 1.5 x ULN.
* Phase 2 only: Active malignancy (except for renal cell carcinoma, melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months.
* Known intolerance to any of the study drugs (or any of the excipients) and/or known hypersensitivity to rapamycins (e.g., sirolimus, everolimus, temsirolimus) or any of the excipients.
* Phase 1b only: Subjects who discontinued prior tyrosine kinase inhibitor due to toxicity will be ineligible.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2014-06-13 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Limited
Locations (37):
- United States (14):
  - Tucson, Arizona
  - Orange, California
  - San Diego, California
  - Tampa, Florida
  - Joliet, Illinois
  - Louisville, Kentucky
  - Annapolis, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Tupelo, Mississippi
  - New York, New York
  - Tulsa, Oklahoma
  - Charleston, South Carolina
  - Dallas, Texas
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Poland (4):
  - Gdansk
  - Lodz
  - Szczecin
  - Warsaw
- Spain (4):
  - Barcelona
  - Córdoba
  - Madrid
  - Pamplona
- United Kingdom (12):
  - Bristol
  - Cambridge
  - Cardiff
  - Glasgow
  - Guildford
  - Ipswich
  - Leicester
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Southampton
  - Surrey

REFERENCES:
- [Derived] Lee CH, Motzer RJ, Glen H, Michaelson MD, Larkin J, Minoshima Y, Kanekiyo M, Ikezawa H, Sachdev P, Dutcus CE, Funahashi Y, Voss MH. Correlative serum biomarker analyses in the phase 2 trial of lenvatinib-plus-everolimus in patients with metastatic renal cell carcinoma. Br J Cancer. 2021 Jan;124(1):237-246. doi: 10.1038/s41416-020-01092-0. Epub 2020 Oct 7. PMID 33024271
- [Derived] Motzer RJ, Hutson TE, Glen H, Michaelson MD, Molina A, Eisen T, Jassem J, Zolnierek J, Maroto JP, Mellado B, Melichar B, Tomasek J, Kremer A, Kim HJ, Wood K, Dutcus C, Larkin J. Lenvatinib, everolimus, and the combination in patients with metastatic renal cell carcinoma: a randomised, phase 2, open-label, multicentre trial. Lancet Oncol. 2015 Nov;16(15):1473-1482. doi: 10.1016/S1470-2045(15)00290-9. Epub 2015 Oct 22. PMID 26482279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 173 participants were enrolled into the study and treated.
Groups:
- Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (12 mg) and everolimus (5 mg) were taken once daily in continuous 28-day cycles. Dose Escalation Cohort-Cycle 1: both study drugs were taken at the same time of day in a fasting state with water. Cycles 2, 3, etc. and Expansion Cohort: both study drugs were taken at the same time of day with water, either after a meal or in a fasting state. Dose escalation began with 3 participants in Cohort 1. If no dose-limiting toxicity (DLT) occurred, then enrollment proceeded to Cohort 2. If 1 participant had a DLT, 3 more participants were enrolled in Cohort 1. If 1 or none of the 6 participants had a DLT, then enrollment proceeded to Cohort 2.
  If 2 or more participants had a DLT during Cycle 1, the dose escalation committee (DEC) decided if they were lenvatinib-related and if enrollment could proceed, lenvatinib was reduced to 6 mg daily (everolimus dose was not reduced). If it could not be determined that the DLTs were lenvatinib-related, enrollment stopped.
- Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (18 mg) and everolimus (5 mg) were taken once daily in continuous 28-day cycles. Dose Escalation Cohort-Cycle 1: both study drugs were taken at the same time of day in the fasting state with water. Cycles 2, 3, etc. and Expansion Cohort: both study drugs were taken at the same time of day with water, either after a meal or in a fasting state. Dose escalation began with 3 participants in Cohort 1. If no DLT occurred, then enrollment would proceed to Cohort 3. If 1 participant had a DLT, 3 more participants were enrolled in Cohort 2. If 1 or none of the 6 participants exhibited a DLT, enrollment proceeded to Cohort 3.
  If 2 or more participants had a DLT during Cycle 1, dose escalation ceased and additional participants were enrolled to the next lower dose to achieve a total of 6 participants in that cohort.
- Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (24 mg) and everolimus (5 mg) were taken once daily in continuous 28-day cycles. Dose Escalation Cohort-Cycle 1: both study drugs were taken at the same time of day in the fasting state with water. Cycles 2, 3, etc. and Expansion Cohort: both study drugs were taken at the same time of day with water, either after a meal or in a fasting state. Dose escalation began with 3 participants in Cohort 1. If no DLT occurred, then enrollment proceeded to Cohort 4. If 1 participant had a DLT, 3 more participants were enrolled Cohort 3. If 1 or none of the 6 participants exhibited a DLT, then enrollment proceeded to Cohort 4.
  If 2 or more participants had a DLT during Cycle 1, dose escalation ceased and additional participants were enrolled to the next lower dose to achieve a total of 6 participants in that cohort.
- Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus: The DLT was achieved and no participants were enrolled into this cohort.
- Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (18mg) and everolimus (5 mg) was once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles. Treatment cycles began with the first dose of study drug in Cycle 1 and continued in 28-day (4-week) consecutive cycles until completion of the off-treatment assessments (within 30 days after the last study treatment administration). Study drugs were administered at the clinic for the first dose and on the pharmacokinetic (PK) sampling days.
- Phase 2 (Arm B): 24 mg Lenvatinib: Oral lenvatinib (24 mg) was taken once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles.
- Phase 2 (Arm C): 10 mg Everolimus: Oral everolimus (10 mg) was taken once daily in the morning (consistently either with or without food) with water, in continuous 28-day (4-week) cycles.
Period: Phase 1b
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Started | 7 (Participants in Phase 1b did not advance to Phase 2.) | 11 (Participants in Phase 1b did not advance to Phase 2.) | 2 (Participants in Phase 1b did not advance to Phase 2.) | 0 (Participants in Phase 1b did not advance to Phase 2.) | 0 | 0 | 0
Completed | 6 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Participant Choice | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative-Withdrew Consent | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Started | 0 | 0 | 0 | 0 | 51 (Participants in Phase 2 did not participate in Phase 1b.) | 52 (Participants in Phase 2 did not participate in Phase 1b.) | 50 (Participants in Phase 2 did not participate in Phase 1b.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 51 | 52 | 50
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 30 | 32 | 38
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 11 | 13 | 5
Not completed — Participant Choice | 0 | 0 | 0 | 0 | 3 | 0 | 1
Not completed — Administrative-Withdrew Consent | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 6 | 7 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (18 mg) and everolimus (5 mg) was once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles. Treatment cycles began with the first dose of study drug in Cycle 1 and continued in 28-day (4-week) consecutive cycles until completion of the off-treatment assessments (within 30 days after the last study treatment administration). Study drugs were administered at the clinic for the first dose and on the pharmacokinetic (PK) sampling days.
- Total: Total of all reporting groups
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus | Total
Number analyzed (Participants) | 7 | 11 | 2 | 0 | 51 | 52 | 50 | 173
Age, Customized [Geometric Mean (Standard Deviation); unit: Years]
  Phase 1b | 58.0 (3.92) | 58.1 (7.97) | 61.0 (2.83) |  | 0 (0) | 0 (0) | 0 (0) | 58.4 (6.29)
  Phase 2 | 0 (0) | 0 (0) | 0 (0) |  | 61.7 (8.2) | 63.3 (8.6) | 58.9 (9.2) | 61.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 |  | 16 | 13 | 12 | 47
  Male | 4 | 9 | 1 |  | 35 | 39 | 38 | 126

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicity (DLT)
Description: A DLT was defined as either a treatment-related failure to administer greater than or equal to (>=) 75% of the planned dosage of lenvatinib/everolimus or a specific National Cancer Institute Common Toxicity Criteria (NCI CTC) >= Grade 3 (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care daily living activities) hematologic or nonhematologic toxicities considered to be possibly related to lenvatinib and/or everolimus therapy assessed during the first treatment cycle of each dose level. Higher grade indicates more severe toxicity.
Time Frame: First dose of study drug (Cycle 1 Day 1) to end of first 4 weeks of therapy (Cycle 1)
Population: Safety analysis set included all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Groups:
- Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (24 mg) and everolimus (5 mg) were taken once daily in continuous 28-day cycles. Dose Escalation Cohort-Cycle 1: both study drugs were taken at the same time of day in the fasting state with water. Cycles 2, 3, etc. and Expansion Cohort: both study drugs were taken at the same time of day with water, either after a meal or in a fasting state. Dose escalation began with 3 participants in Cohort 1. If no DLT occurred, then enrollment would proceed to Cohort 3. If 1 participant had a DLT, 3 more participants were enrolled in Cohort 2. If 1 or none of the 6 participants exhibited a DLT, enrollment proceeded to Cohort 3.
  If 2 or more participants had a DLT during Cycle 1, dose escalation ceased and additional participants were enrolled to the next lower dose to achieve a total of 6 participants in that cohort.
- Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (18 mg) and everolimus (5 mg) were taken once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles. Treatment cycles began with the first dose of study drug in Cycle 1 and continued in 28-day (4-week) consecutive cycles until completion of the off-treatment assessments (within 30 days after the last study treatment administration). Study drugs were administered at the clinic for the first dose and on the pharmacokinetic (PK) sampling days.
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 7 | 11 | 2 | 0 | 0 | 0 | 0
Participants
  Grade 3 abdominal pain | 1 | 0 | 0 |  |  |  |
  Grade 2 fatigue with Grade 1 GI reflux & anorexia | 0 | 1 | 0 |  |  |  |
  Grade 3 nausea | 0 | 0 | 1 |  |  |  |
  Grade 2 stomatitis | 0 | 0 | 1 |  |  |  |

2. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) and Recommended Phase 2 (RP2) Dose
Description: The highest dose level resulting in 0 or 1 DLT in 6 participants was to be considered the MTD of Phase 1b. Once the MTD was established, the participant cohort was expanded to a minimum of 10 participants. The MTD was confirmed by assessing DLTs during Cycle 1 and intolerable toxicities (i.e., not manageable with dose interruption and/or reduction) during Cycle 2 of therapy. Once the dose of lenvatinib/everolimus combination to be used in the succeeding Phase 2 part of the study was established, enrollment into Phase 2 was started. The RP2 dose was the same as the confirmed MTD and was used for the Phase 2 Treatment Arm A of this study.
Time Frame: First dose of study drug (Cycle 1 Day 1) to end of Cycle 2 (1 cycle = 28 days/4 weeks)
Population: Safety analysis set included all participants who received at least one dose of study treatment.
Measure: Number; unit: mg/day
Groups:
- Phase 1b: Dose Escalation and MTD Expansion Cohorts: Oral everolimus (18 mg) and lenvatinib (5 mg) were taken once daily in the morning (consistently with or without food) with water. Any dietary habits around the time of study medication intake had to be kept as consistent as possible throughout the study.
Arm/Group | Phase 1b: Dose Escalation and MTD Expansion Cohorts
Number analyzed (Participants) | 11
mg/day | 18.0

3. Primary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS was defined as the time (in months) from the date of first dose of study drug to the first documentation of disease progression or death, whichever occurred first. Kaplan-Meier (K-M) estimates were used to estimate median PFS, presented with 2-sided 95% confidence intervals (CIs). Tumor assessments were performed every 8 weeks (or sooner if there was evidence of progressive disease using computed tomography (CT) or magnetic resonance imaging (MRI) and scan acquisition techniques (including use or nonuse of intravenous (IV) contrast). Tumor response was determined at the site by the investigator and radiologist using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 in the evaluation of the tumor assessment scans. The date of objective disease progression was defined as the earliest date of radiological disease progression. Participants removed from therapy due to clinical progression with no radiologic confirmation were censored at their last radiologic assessment date.
Time Frame: Date of randomization into Phase 2 (Cycle 1 Day 1) to the date of first documentation of disease progression or death (whichever occurred first), assessed up to data cutoff date (13 Jun 2014), up to approximately 2 years and 3 months
Population: Full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 52 | 50
Months |  |  |  |  | 14.6 [5.9 to 20.1] | 7.4 [5.6 to 10.2] | 5.5 [3.5 to 7.1]
Statistical Analysis 1: Comparison: Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus vs Phase 2 (Arm C): 10 mg Everolimus; Null hypothesis of no difference in PFS was analyzed using the stratified log-rank test with hemoglobin (less than or equal to 13 g/dL vs greater than 13 g/dL for males; and less than or equal to 11.5 g/dL vs greater than 11.5 g/dL for females) and corrected serum calcium (greater than or equal to 10 mg/dL vs less than 10 mg/dL) as stratification factors. Each null hypothesis was tested at a nominal alpha=0.05; Test type: Superiority or Other; p = 0.0005, Log Rank; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.24 to 0.68] — Hazard ratio between treatment groups and corresponding 95% CI was estimated using the stratified Cox regression model (stratified by hemoglobin and corrected serum calcium) with treatment as a factor
Statistical Analysis 2: Comparison: Phase 2 (Arm B): 24 mg Lenvatinib vs Phase 2 (Arm C): 10 mg Everolimus; Test type: Superiority or Other; p = 0.0479, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.38 to 0.98]
Statistical Analysis 3: Comparison: Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus vs Phase 2 (Arm B): 24 mg Lenvatinib; Test type: Superiority or Other; p = 0.1209, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.39 to 1.10]

4. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization until date of death from any cause. Median survival time was calculated using K-M estimate for each treatment arm and presented with 2-sided 95% CIs. Participants who were lost to follow-up or alive at the data cutoff date (10 Dec 2014) were censored at the date the participants were last known to be alive.
Time Frame: Randomization (Cycle 1 Day 1) until date of death from any cause, assessed up to the data cutoff date (10 Dec 2014), up to approximately 2 years and 9 months
Population: Full analysis set which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 52 | 50
Months |  |  |  |  | 25.5 [16.4 to NA] — NA = not estimable | 19.1 [13.6 to 26.2] | 15.4 [11.8 to 19.6]
Statistical Analysis 1: Comparison: Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus vs Phase 2 (Arm C): 10 mg Everolimus; Planned analyses were performed to test null hypothesis of treatment difference in OS at a nominal significance level of 0.05 (2-sided) using the stratified log-rank test using stratification factors; Test type: Superiority or Other; p = 0.0242, Log Rank; Hazard Ratio (HR) = 0.514, 95% CI 2-sided [0.299 to 0.884] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 2 (Arm B): 24 mg Lenvatinib vs Phase 2 (Arm C): 10 mg Everolimus; Test type: Superiority or Other; p = 0.1181, Log Rank; Hazard Ratio (HR) = 0.684, 95% CI 2-sided [0.411 to 1.138]
Statistical Analysis 3: Comparison: Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus vs Phase 2 (Arm B): 24 mg Lenvatinib; Test type: Superiority or Other; p = 0.3157, Log Rank; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.433 to 1.301]

5. Secondary Outcome: Phase 2: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants who had the best overall response (BOR) of complete response (CR) or partial response (PR) as determined by the investigator, using RECIST 1.1 in the evaluation of MRI or CT scans of targeted lesions. Tumor assessments were performed every 8 weeks (or sooner if there was evidence of progressive disease). The BOR was defined as the best response recorded from the start of the study treatment until discontinuation from the study. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR was calculated with exact 95% CIs using the method of Clopper and Pearson.
Time Frame: Randomization (Cycle 1 Day 1) until first evidence of disease progression, assessed up to the data cutoff date (13 Jun 2014), or up to approximately 2 years and 3 months
Population: Full analysis set which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 52 | 50
Percentage of participants |  |  |  |  | 43.1 [29.3 to 57.8] | 26.9 [15.6 to 41.0] | 6.0 [1.3 to 16.5]
Statistical Analysis 1: Comparison: Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus vs Phase 2 (Arm C): 10 mg Everolimus; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Analysis performed after database lock. P-value was based on the 2-sided Fisher's exact P-value; Rate ratio = 7.2, 95% CI 2-sided [2.3 to 22.5] — Rate ratio was based on the normal approximation
Statistical Analysis 2: Comparison: Phase 2 (Arm B): 24 mg Lenvatinib vs Phase 2 (Arm C): 10 mg Everolimus; Test type: Superiority or Other; p = 0.0067, Fisher Exact — Analysis performed after database lock. P-value was based on the 2-sided Fisher's exact P-value; Rate ratio = 4.5, 95% CI 2-sided [1.4 to 14.7]
Statistical Analysis 3: Comparison: Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus vs Phase 2 (Arm B): 24 mg Lenvatinib; Test type: Superiority or Other; p = 0.1007, Fisher Exact — Analysis performed after database lock. P-value was based on the 2-sided Fisher's exact P-value; Rate ratio = 1.6, 95% CI 2-sided [0.9 to 2.8]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who had a BOR of CR or PR or SD (minimum duration from randomization to SD greater than or equal to 7 weeks). Assessments were performed every 8 weeks and were based on investigator review data using RECIST 1.1. The 95% CI was constructed using the method of Clopper and Pearson. DCR = CR + PR + SD greater than or equal to 7 weeks.
Time Frame: Baseline (Randomization) to first evidence of disease progression, assessed up to the data cutoff date (13 Jun 2014), or up to approximately 2 years and 3 months
Population: Full analysis set which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (12 mg) and everolimus (5 mg) were taken once daily in continuous 28-day cycles. Dose Escalation Cohort-Cycle 1: both study drugs were taken at the same time of day in a fasting state with water. Cycles 2, 3, etc. and Expansion Cohort: both study drugs were taken at the same time of day withwater, either after a meal or in a fasting state. Dose escalation began with 3 participants in Cohort 1. If no dose-limiting toxicity (DLT) occurred, then enrollment proceeded to Cohort 2. If 1 participant had a DLT, 3 more participants were enrolled in Cohort 1. If 1 or none of the 6 participants had a DLT, then enrollment proceeded to Cohort 2.
  If 2 or more participants had a DLT during Cycle 1, the dose escalation committee (DEC) decided if they were lenvatinib-related and if enrollment could proceed, lenvatinib was reduced to 6 mg daily (everolimus dose was not reduced). If it could not be determined that the DLTs were lenvatinib-related, enrollment stopped.
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 52 | 50
Percentage of participants |  |  |  |  | 84.3 [71.4 to 93.0] | 78.8 [65.3 to 88.9] | 68.0 [53.3 to 80.5]

7. Secondary Outcome: Durable Stable Disease (SD) Rate
Description: The durable SD rate was defined as the percentage of participants whose BOR was SD and the duration of SD was greater than or equal to 23 weeks. The durable SD was based on investigator review data using RECIST 1.1. The 95% CI was constructed using the method of Clopper and Pearson.
Time Frame: as for outcome 6
Population: Full analysis set which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 52 | 50
Percentage of participants |  |  |  |  | 25.5 [14.3 to 39.6] | 38.5 [25.3 to 53.0] | 36.0 [22.9 to 50.8]

8. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants who had BOR of CR, PR, or durable SD (duration of SD was greater than or equal to 23 weeks) and was based on investigator review data using RECIST 1.1. The BOR was defined as the best response recorded from the start of study treatment until discontinuation from the study. There was no requirement for confirmatory measurement of PR or CR to deem either one the BOR. The 95% CI was constructed using the method of Clopper and Pearson. CBR = CR + PR + SD greater than or equal to 23 weeks.
Time Frame: as for outcome 6
Population: Full analysis set which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2 (Arm C): 10 mg Everolimus: Oral everolimus (10 mg) was taken once daily in the morning (consistently either with or without food) with water, in continuous 28-day (4 week) cycles.
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 52 | 50
Percentage of participants |  |  |  |  | 68.6 [54.1 to 80.9] | 65.4 [50.9 to 78.0] | 42.0 [28.2 to 56.8]

9. Secondary Outcome: Summary of Plasma Concentrations of Lenvatinib for Sparse Pharmacokinetic (PK) Sampling for Phase 1b and Phase 2
Description: Blood samples were collected during the Randomization Phase. Most participants had 6 samples taken over 3 cycles of treatment (sparse sampling - 2 samples taken per cycle, one at predose and one at 2 to 8 hours postdose). Plasma concentrations of lenvatinib were measured and concentration data were summarized. The summary statistics at time points with one or more below the limit of quantitation (BLQ) values were calculated by assigning zero for each BLQ value.
Time Frame: Cycle 1 (Day 1), Cycle 2 (Day 1), Cycle 3 (Day 1)
Population: Pharmacokinetic analysis set included all participants who have received at least one dose of study drug (lenvatinib or everolimus) and have evaluable concentration data.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Cycle 1, Day 1 (0 Hours); Cycle 2, Day 1 (0 Hours); Cycle 3, Day 1 (0 Hours): Lenvatinib (18 mg) and everolimus (5 mg) were administered as described previously. Blood samples were collected immediately prior to study drug administration.
- Cycle 1, Day 1 (2-8 Hours); Cycle 2, Day 1 (2-8 Hours); Cycle 3, Day 1 (2-8 Hours): Lenvatinib (18 mg) and everolimus (5 mg) were administered as described previously. Blood samples were collected 2 to 8 hours after study drug administration.
Arm/Group | Cycle 1, Day 1 (0 Hours) | Cycle 1, Day 1 (2-8 Hours) | Cycle 2, Day 1 (0 Hours) | Cycle 2, Day 1 (2-8 Hours) | Cycle 3, Day 1 (0 Hours) | Cycle 3, Day 1 (2-8 Hours)
Number analyzed (Participants) | 57 | 55 | 45 | 41 | 42 | 40
ng/mL | 5.6 (29.8) | 197 (140) | 66.9 (52.7) | 237 (154) | 37.0 (35.5) | 180 (118)

10. Secondary Outcome: Summary of Blood Concentrations of Everolimus for Sparse PK Sampling for Phase 1b and Phase 2
Description: Blood samples were collected during the Randomization Phase. Most participants had 6 samples taken over 3 cycles of treatment (sparse sampling - 2 samples taken per cycle, one at predose and one at 2 to 8 hours postdose). Whole blood concentrations of everolimus were measured and concentration data were summarized. The summary statistics at time points with one or more BLQ values were calculated by assigning zero for each BLQ value.
Time Frame: Cycle 1 (Day 1), Cycle 2 (Day 1), Cycle 3 (Day 1)
Population: Pharmacokinetic analysis set included all participants who received at least one dose of study drug (lenvatinib or everolimus) and had evaluable concentration data.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cycle 1, Day 1 (0 Hours) | Cycle 1, Day 1 (2-8 Hours) | Cycle 2, Day 1 (0 Hours) | Cycle 2, Day 1 (2-8 Hours) | Cycle 3, Day 1 (0 Hours) | Cycle 3, Day 1 (2-8 Hours)
Number analyzed (Participants) | 37 | 35 | 29 | 28 | 27 | 25
ng/mL | 0.0 (0.00) | 19.4 (9.16) | 10.0 (7.28) | 24.3 (14.2) | 6.8 (6.06) | 26.4 (14.8)

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC(0-24)) for Lenvatinib When Administered Alone or in Combination With Everolimus
Description: Between 9 and 12 participants in each of the 3 treatment arms participated in an optional substudy where instead of the sparse sampling, 9 samples were to be taken over 1 single 24-hour period (i.e., intensive sampling) for full PK profiling. Blood samples were analyzed for study drug using standardized methods. PK parameters for lenvatinib were derived from lenvatinib concentration data using non-compartmental methods. Data were compared via descriptive statistics between single agent and combination therapy.
Time Frame: Phase 2: Cycle 1 Day 15 immediately predose, and 30 minutes, 1, 2, 3, 4, 8, 12 (optional), and 24 hours postdose (predose on Day 16)
Population: Pharmacokinetic sub analysis set consisted of all participants who agreed to participate in the intensive PK sampling portion of Phase 2 of the study, had received at least 1 dose of study drug (lenvatinib or everolimus), and had evaluable concentration data.
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Groups:
- Phase 2: 18 mg Lenvatinib + 5 mg Everolimus: Oral lenvatinib (18mg) and everolimus (5 mg) were taken once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles. Treatment cycles began with the first dose of study drug in Cycle 1 and continued in 28-day (4-week) consecutive cycles until completion of the off-treatment assessments (within 30 days after the last study treatment administration). Study drugs were administered at the clinic for the first dose and on the pharmacokinetic (PK) sampling days.
- Phase 2: 24 mg Lenvatinib: Oral lenvatinib (24 mg) was taken once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles.
Arm/Group | Phase 2: 18 mg Lenvatinib + 5 mg Everolimus | Phase 2: 24 mg Lenvatinib
Number analyzed (Participants) | 8 | 9
ng·hr/mL | 3185 (1030) | 5252 (2717)

12. Secondary Outcome: Maximum Concentration (Cmax) of Lenvatinib in Plasma When Administered Alone or in Combination With Everolimus
Description: Cmax for lenvatinib was defined as the maximum observed concentration of lenvatinib in plasma following administration of study treatment on Cycle 1 Day 15 and was obtained directly from the measured plasma concentration-time curves.
Time Frame: Phase 2: Cycle 1 Day 15
Population: PK sub analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: 18 mg Lenvatinib + 5 mg Everolimus | Phase 2: 24 mg Lenvatinib
Number analyzed (Participants) | 8 | 9
ng/mL | 327 (179) | 403 (165)

13. Secondary Outcome: Time to Cmax (Tmax) for Lenvatinib When Administered Alone or in Combination With Everolimus
Description: Tmax for lenvatinib was the amount of time taken after administration of study treatment on Cycle 1 Day 15 to reach maximum concentration (Cmax) of lenvatinib in plasma.
Time Frame: Phase 2: Cycle 1 Day 15
Population: PK sub analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 2: 18 mg Lenvatinib + 5 mg Everolimus | Phase 2: 24 mg Lenvatinib
Number analyzed (Participants) | 8 | 9
Hours | 2.0 [2.0 to 8.2] | 4.0 [0.5 to 8.0]

14. Secondary Outcome: Area Under the Blood Concentration-Time Curve From 0 to 24 Hours for Everolimus When Administered Alone or in Combination With Lenvatinib
Description: Between 9 and 12 participants in each of the 3 treatment arms participated in an optional substudy where instead of the sparse sampling, 9 samples were to be taken over 1 single 24-hour period (i.e., intensive sampling) for full PK profiling. Blood samples were analyzed for study drug using standardized methods. PK parameters for everolimus were derived from everolimus concentration data using non-compartmental methods. Data were compared via descriptive statistics between single agent and combination therapy.
Time Frame: as for outcome 11
Population: PK sub analysis set. n=8 for AUC(0-24)
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Groups:
- Phase 2: 18 mg Lenvatinib + 5 mg Everolimus: Oral lenvatinib (18 mg) and everolimus (5 mg) were taken once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles. Treatment cycles began with the first dose of study drug in Cycle 1 and continued in 28-day (4-week) consecutive cycles until completion of the off-treatment assessments (within 30 days after the last study treatment administration). Study drugs were administered at the clinic for the first dose and on the pharmacokinetic (PK) sampling days.
- Phase 2: 10 mg Everolimus: Oral everolimus (10 mg) was taken once daily in the morning (consistently either with or without food) with water, in continuous 28-day (4-week) cycles.
Arm/Group | Phase 2: 18 mg Lenvatinib + 5 mg Everolimus | Phase 2: 10 mg Everolimus
Number analyzed (Participants) | 4 | 8
ng·hr/mL | 378 (88.1) | 463 (263)

15. Secondary Outcome: Maximum Concentration of Everolimus (Cmax) in Blood When Administered Alone or in Combination With Lenvatinib
Description: Cmax for everolimus was defined as the maximum observed concentration of everolimus in blood following administration of study treatment on Cycle 1 Day 15 and was obtained directly from the measured blood concentration-time curves.
Time Frame: Phase 2: Cycle 1 Day 15
Population: PK sub analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: 18 mg Lenvatinib + 5 mg Everolimus | Phase 2: 10 mg Everolimus
Number analyzed (Participants) | 4 | 11
ng/mL | 38 (14.5) | 54 (24.9)

16. Secondary Outcome: Time to Cmax (Tmax) for Everolimus When Administered Alone or in Combination With Lenvatinib
Description: Tmax for everolimus was the amount of time taken after administration of study treatment on Cycle 1 Day 15 to reach the maximum concentration (Cmax) of everolimus in blood.
Time Frame: Phase 2: Cycle 1 Day 15
Population: PK sub analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 2: 18 mg Lenvatinib + 5 mg Everolimus | Phase 2: 10 mg Everolimus
Number analyzed (Participants) | 4 | 11
Hours | 1.0 [0.5 to 8.0] | 1.0 [0.5 to 25.9]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were collected and defined as those AEs that occurred after the first dose of study medication and up to 30 days after the last dose of study medication. AEs were collected for approximately 4 years.
Description: Safety analysis set included all participants who received at least one dose of study drug/s and had at least one postbaseline safety evaluation. AE severity was assessed using Common Terminology for Adverse Events (CTCAE). Serious AEs were followed until the event resolved or the event or sequelae stabilized.
Groups:
- Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus: Oral lenvatinib (18mg) and everolimus (5 mg) were taken once daily in the morning (consistently with or without food) with water, in continuous 28-day (4-week) cycles. Treatment cycles began with the first dose of study drug in Cycle 1 and continued in 28-day (4-week) consecutive cycles until completion of the off-treatment assessments (within 30 days after the last study treatment administration). Study drugs were administered at the clinic for the first dose and on the pharmacokinetic (PK) sampling days.
Arm/Group | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus | Phase 2 (Arm B): 24 mg Lenvatinib | Phase 2 (Arm C): 10 mg Everolimus
All-Cause Mortality (participants affected / at risk) | 6/7 | 9/11 | 0/2 | 0/0 | 43/51 | 40/52 | 45/50
Serious Adverse Events (participants affected / at risk) | 6/7 | 8/11 | 0/2 | 0/0 | 30/51 | 28/52 | 21/50
Other Adverse Events (participants affected / at risk) | 7/7 | 11/11 | 2/2 | 0/0 | 51/51 | 51/52 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus (N=7) | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus (N=11) | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus (N=2) | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus (N=0) | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus (N=51) | Phase 2 (Arm B): 24 mg Lenvatinib (N=52) | Phase 2 (Arm C): 10 mg Everolimus (N=50)
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection Fraction Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 4 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 3 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 4
Sideroblastic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic Foot Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infectious Pleural Effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Rectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatinine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body Temperature Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram Repolarisation Abnormality (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibrin D Dimer Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carotid Artery Occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (Cohort 1): 12 mg Lenvatinib Plus 5 mg Everolimus (N=7) | Phase 1b (Cohort 2): 18 mg Lenvatinib Plus 5 mg Everolimus (N=11) | Phase 1b (Cohort 3): 24 mg Lenvatinib Plus 5 mg Everolimus (N=2) | Phase 1b (Cohort 4): 24 mg Lenvatinib Plus 10 mg Everolimus (N=0) | Phase 2 (Arm A): 18 mg Lenvatinib Plus 5 mg Everolimus (N=51) | Phase 2 (Arm B): 24 mg Lenvatinib (N=52) | Phase 2 (Arm C): 10 mg Everolimus (N=50)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 7 | 3 | 11
Haemorrhagic Disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 5 | 1 | 4
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Ventricular Hypokinesia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 3 | 0 | 0 | 12 | 19 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye Swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 12 | 11 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 8 | 7 | 3
Anal Pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 6 | 19 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 1 | 0 | 43 | 37 | 17
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 6 | 6 | 6
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 4 | 3 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 0
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Lip Discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 6 | 1 | 0 | 22 | 32 | 8
Oral Mucosal Blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 6 | 5 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 7 | 2 | 0 | 15 | 13 | 21
Vomiting (Gastrointestinal disorders) | 5 | 5 | 1 | 0 | 24 | 20 | 6
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 13 | 8 | 3
Chills (General disorders) | 0 | 2 | 0 | 0 | 2 | 3 | 1
Fatigue (General disorders) | 4 | 11 | 2 | 0 | 26 | 21 | 16
Gait Disturbance (General disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1
Localised Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 1
Oedema Peripheral (General disorders) | 1 | 6 | 0 | 0 | 15 | 9 | 9
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 9 | 5 | 5
Dilatation Intrahepatic Duct Acquired (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 4 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infectious Pleural Effusion (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Lymph Gland Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 7 | 4 | 7
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 3
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 4 | 7 | 7
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 4 | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Periorbital Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 5 | 3 | 3
Amylase Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 2 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1 | 0 | 0 | 2 | 1 | 2
Blood Bilirubin Increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Blood Cholesterol Increased (Investigations) | 0 | 1 | 0 | 0 | 4 | 2 | 3
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2 | 0 | 0 | 4 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Blood Phosphorus Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Blood Potassium Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 2 | 1
Cardiac Murmur (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Computerised Tomogram Thorax Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection Fraction Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Haemoglobin Decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 2 | 5
Lipase Increased (Investigations) | 0 | 2 | 0 | 0 | 4 | 5 | 3
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Murphy's Sign Positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein Urine Present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 2 | 5 | 0 | 0 | 16 | 26 | 4
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 6 | 1 | 0 | 27 | 30 | 10
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 18 | 6 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 8 | 3 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 3 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 7 | 0 | 0 | 18 | 7 | 12
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0 | 14 | 13 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 0 | 11 | 11 | 7
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2 | 2 | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 8 | 7 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 4 | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 4 | 7 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 6 | 6 | 3
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance In Attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 1 | 0 | 2 | 4 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 4 | 4 | 1
Headache (Nervous system disorders) | 4 | 3 | 0 | 0 | 10 | 13 | 4
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 4 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 3 | 1
Confusional State (Psychiatric disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 10 | 8 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 3
Proteinuria (Renal and urinary disorders) | 5 | 6 | 0 | 0 | 13 | 16 | 7
Renal Failure Acute (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Mass (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0 | 0 | 20 | 9 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 10 | 19 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1 | 0 | 11 | 11 | 11
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 4 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 0 | 9 | 4 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 2
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 4 | 2 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 5 | 3 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 4 | 8 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 7 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 0 | 9 | 8 | 11
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2 | 3 | 4
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 5
Skin Mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1
Aortic Dilatation (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypertension (Vascular disorders) | 5 | 4 | 0 | 0 | 21 | 26 | 5
Hypotension (Vascular disorders) | 1 | 3 | 0 | 0 | 3 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 3 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 5
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 0 | 0 | 7 | 2 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 4 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 7 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 3
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 4 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 4 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 7 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Peripheral Swelling (General disorders) | 1 | 1 | 0 | 0 | 5 | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No